CLINICAL TRIAL: NCT01020071
Title: Prospective Evaluation of the Efficacy of Pascal Laser Iridotomy and Pascal Laser Peripheral Iridoplasty: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Ophthalmology, Associate Professor Paul Chew, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB A/09/93
Record Dates: First submitted 2009-11-22; First posted 2009-11-25 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Glaucoma
Keywords: iridotomy; iridoplasty; angle closure glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Angle-Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- laser treatment (Other): laser peripheral iridotomy and laser peripheral iridoplasty
  Interventions: Procedure: pattern scanning laser iridotomy and iridoplasty

INTERVENTIONS:
Procedure: pattern scanning laser iridotomy and iridoplasty — peripheral laser iridotomy and iridoplasty using pattern scanning laser technique
  Other Names: PASCAL

SUMMARY:
Objective: The main objective of this study is to evaluate the efficacy of Pascal Laser Iridotomy and Pascal Laser Peripheral Iridoplasty in lowering intraocular pressure and opening up the angles in patients with narrow angles, primary angle closure and primary angle closure glaucoma.

The specific objectives are to evaluate the pain and inflammation associated with the procedure and its possible adverse effects on the lens and corneal endothelium.

Study Design: Prospective, interventional case series Study Population: Healthy males and females with appositional angle closure aged 21 y/o and above Methods: Potential participants are evaluated by a glaucoma specialist in National University Hospital. If they are identified as having appositional angle closure they are invited to participate in the study and assigned to either iridotomy or iridoplasty depending on the mechanism of angle closure present. Pupil block for Pascal Laser Iridotomy and plateau iris and angle crowding for Pascal Laser Peripheral Iridoplasty. If they agree to participate they will undergo visual acuity, slit lamp examination, intraocular pressure determination by Goldmann Applanation Tonometry, gonioscopy, optic nerve head evaluation by indirect ophthalmoscopy and lens evaluation by LOCS III opacity grading system. Humphrey visual field examination using 24-2 SITA standard algorithm and stereodisc photos will be obtained if not done within the past 12 months. Anterior segment OCT and laser flare meter will also be performed prior to the procedure. Enrolled patients will be divided into 2 groups. The first group will be assigned to Pascal Laser Iridotomy. The primary mechanism of angle closure in this group is pupillary block. The second group will be assigned to Pascal Laser Peripheral Iridoplasty. This group has non-pupil bock mechanisms which include plateau iris or angle crowding. After the laser procedure, follow-up examinations will be done 1 hr post laser, 1 week, 1 month, 3 months and 6 months.

Outcome Measures: The primary outcome measures are the intraocular pressure difference pre and post laser and the opening of angles. Secondary outcome measures are pain and inflammation associated with laser procedure, lens and corneal endothelial changes.

DETAILED DESCRIPTION:
PLANNED INTERVENTIONS Potential study participants are seen by a glaucoma specialist at National University Hospital. If they are identified as having primary angle closure and have met the inclusion criteria mentioned above, they will be invited to participate in the study. Potential risks and benefits will be explained. After which, they will sign an informed consent when they agree to participate.

Visual acuity, slit lamp examination, intraocular pressure determination through Goldmann Applanation Tonometry, gonioscopy, optic nerve head examination through indirect ophthalmoscopy and lens evaluation using LOCS III lens opacity grading system will be done on baseline visit. Humphrey visual field exam using 24-2, SITA standard algorithm and stereodisc photos will also be obtained if not done within the past 12 months. Anterior segment OCT, laser flare meter of the anterior chamber and corneal endothelial cell count will also be done.

Based on gonioscopy and anterior segment OCT findings, the primary mechanism of angle closure will be analyzed. Depending on the major mechanism, they will be assigned to either Pascal Laser Iridotomy and Pascal Laser Peripheral Iridoplasty. Patients identified as having pupil block will be assigned to Pascal Laser Iridotomy and those identified as having plateau iris configuration, plateau iris syndrome or angle crowding will be assigned to Pascal Laser Peripheral Iridoplasty.

Post laser follow up will be done after 1 week, 1 month, 3 months and 6 months.

PASCAL LASER IRIDOTOMY Prior to laser procedure 1 drop each of Alphagan-P and 4% Pilocarpine are instilled 15 minutes prior.

A. Scanning Laser Parameters

1. Set the pattern mode to square array, 2 x 2 spots, 0.25 distance between spots.
2. Set pulse duration to 20 ms
3. Adjust spot size to 100 um.
4. Apply spots to peripheral iris preferably in the area between 11:00 and 1:00 o'clock position, positioning within an iris crypt until there is thinning of the iris stroma with a honeycomb apearance is obtained. The desired result is the appearance of a small hole with a dark brown base at the base of the burn and dispersion of debris into anterior chamber.

B. Penetrating Burn with Yag Laser

1. Set power to 2-3 mJ
2. Apply laser burns to center of the hole until a mushroom cloud admixed with aqueous balloons into the anterior chamber.
3. Enlarge the hole until approximately 300 um or more.

C. Lens: Abraham lens

PASCAL LASER PERIPHERAL IRIDOPLASTY Prior to laser procedure 1 drop each of Alphagan-P and 4% Pilocarpine are instilled 15 minutes prior.

A. Titrate Average Laser Power

1. Set the pattern mode to single spot
2. Set the pulse duration to 100 ms
3. Adjust spot size to 100 um
4. Apply spots at the peripheral iris one at a time while increasing average power until adequate contraction of peripheral iris is seen.

B. Scanning Laser Parameters

1. Choose the number of rows of spots (2-4) depending on dose.
2. Choose spot separation between arcs from -0.25 to 0.25 spot diameter. One spot diameter = 100 um.
3. Choose spot spacing within each arc from 0 to 1 spot diameter depending on dose.
4. Set radius of the arc to match the curvature of the peripheral iris.

C. Contact lens: CGIL lens

Treat 360 degrees of peripheral iris with a total of 20-24 burns.

DEFINITION OF OUTCOMES The main outcome measures are the difference in the pre laser and post laser intraocular pressures and the opening of angles documented by gonioscopy and anterior segment OCT.

Secondary outcome measures are the pain and inflammation associated with the procedure as seen through slit lamp examination grading of anterior chamber cells and flares and laser flare meter analysis, and the possible changes in the corneal endothelium as seen in the specular microscopy.

Details of Examination Procedures:

1. Visual Acuity Visual acuity: This will be assessed using a logMAR chart under standard lighting: best corrected visual acuity will be recorded (using the subjective refractive correction obtained above). Subjects will start reading at the 6/12 equivalent line (0.3) and if unable to read at least three letters, they will begin to read the line above and continue this process until at least three letters on one line have been read. This line will be recorded as the visual acuity. If the subject is able to read at least three letters on the first line, they will proceed on to the next line below, until they are unable to read further down the chart. If unable to read the chart at 4 m, the subject will be moved to 2m, and then 1m from the chart. If unable to see/achieve minimum recordable logMAR acuity, the vision will be recorded as perception or non-perception of light.
2. Goldman Applanation Tonometry The IOP will be measured by Goldman Applanation Tonometry after instillation of a topical anesthetic. The IOP at every visit will be taken using the same slit lamp and tonometer. Three consecutive readings will be taken and the mean of the three values used in the statistical analyses.
3. Slit lamp Biomicroscopic Examination Slit lamp biomicroscopic examination will be performed on the same slit lamp every visit. Examination of the conjunctiva, cornea, anterior chamber and lens will be done and any abnormalities noted. The lens will be graded using the Lens Opacity Classification Scale III (LOCS III). The anterior cells and flares will be graded as follows: A parallelepiped about 2 mm wide and 4 mm high at 45 degrees will be directed into the pupil. The following table will be used9.

   Grade Aqueous Cells Grade Flare 0 None 0 Complete absence 1 5-10 cells per field 1 Faint flare (barely detectable) 2 10-20 per field 2 Moderate flare (iris and lens details clear) 3 20-50 cells per field 3 Marked flare (iris and lens details hazy) 4 50 + cells per field 4 Intense flare (fixed, coagulated aqueous humor with considerable fibrin)
4. Gonioscopy Gonioscopy will be performed on all patients using Sussman 4-mirror gonioscopy lens to facilitate indentation gonioscopy. Findings in each quadrant will be graded using the Shaffer System and recorded in a goniogram.
5. LOCS III Lens Opacity Grading System LOCS III lens opacity grading system will be used to assess if there will be developing cataract or increasing degree of cataract associated with the laser procedure. It will be done on the baseline visit as well on all follow-up visits.
6. Visual Field Testing Humphrey Visual field Analyzer will be used with the program of SITA standard, 24-2 test. For the visual fields to be reliable, the following criteria should be followed: fixation losses of less than 33%, false positive errors of less than 20% and false negative errors of less than 20%. Mean deviation and pattern standard deviation will be compared on each test to determine progression of the disease.
7. Anterior Segment OCT Anterior segment OCT using Carl Zeiss Visante is an non-contact imaging system used to assess the anterior chamber anatomy especially the anterior chamber angles. It will be performed prelaser, 1 week, 1 month, 3 months and 6 months post laser.
8. Flare Meter The Kowa FM-600 Laser flare meter will be used to assess anterior chamber inflammation. Five measurements will be taken and the average will be recorded as the correct value. Results will be expressed in photons/ms.
9. Corneal Specular Microscopy Non-contact specular microscopy will be performed at the central and peripheral regions of the cornea using Topcon SP-2000P.

This method measures the state of the corneal endothelium, the parameters to be determined are endothelial cell density, cell area, coefficient of variation (CV) in cell area and hexagonality.

SCHEDULE OF STUDY VISITS Recruitment visit Baseline assessment will be done upon referral for inclusion in the study.

Treatment Visit Pascal Laser Iridotomy or Pascal Laser Peripheral Iridoplasty will be done.

Follow-up Visits Follow-up examinations will be performed 1 week, 1 month, 3 months and 6 months after the laser procedure. The following examinations will be done on each postlaser visit: visual acuity, slit lamp examination, intraocular pressure determination, lens opacity evaluation, gonioscopy, anterior segment OCT, laser flare meter examination of anterior chamber inflammation, Humphrey visual fields(baseline & six months) and corneal endothelial cell count.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females having 2 sighted eyes aging 21 y/o and above
* primary angle closure with pupil block component
* plateau iris syndrome or plateau iris configuration
* occludable angles 180 deg and above
* have uncontrolled IOP (>21 mmHg)
* able to follow up
* able to give informed consent

Exclusion Criteria:

* advanced visual field defect affecting 10 degrees of fixation
* previous ocular surgeries
* advanced corneal edema or opacification
* flat anterior chamber
* synechially closed angles
* coexisting ocular pathology except cataract

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are the intraocular pressure difference pre and post laser and the opening of angles. | 6 months

SECONDARY OUTCOMES:
Secondary outcome measures are pain and inflammation associated with laser procedure, lens and corneal endothelial changes. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul TK Chew, FRCOphth, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Kent Ridge, Singapore, Singapore